CLINICAL TRIAL: NCT03472001
Title: Effects of Structured Reflection and Immediate Feedback in Improving of Medical Students' Evaluation of Skin Lesions
Brief Title: Reflection and Feedback in Clinical Reasoning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Hyun-Sun Yoon, Clinical professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SMG-180105
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training group (Experimental): 2-hour training based on reflection and feedback
  Interventions: Other: Reflection and feedback
- Lecture group (Active Comparator): 1-hour lecture
  Interventions: Other: Lecture
- Control group (No Intervention): The remaining students only attending dermatology electives

INTERVENTIONS:
Other: Reflection and feedback — 2-hour training involving 10 written clinical cases to encourage students to practice thinking like a dermatologist in their clinical reasoning, and to help students build adequate illness scripts of skin diseases
  Arms: Training group
Other: Lecture — Traditional didactic lecture which uses the same clinical cases
  Arms: Lecture group

SUMMARY:
Medical students' abilities to diagnose skin lesions after dermatology electives often remain unsatisfactory despite a dermatology elective being one of the most effective ways to improve their clinical reasoning. Feedback and reflection are two basic teaching methods used in clinical settings. This study aimed to investigate the effectiveness of structured reflection and immediate feedback in improving of medical students' evaluation of skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* Fourth-year medical students at Seoul National University College of Medicine
* Students taking 2-week dermatology elective courses

Exclusion Criteria:

* Students who do not complete the whole course

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy in the training set | At the end of a 2-week dermatology elective
  Mean score of the training set (number of correct answers)

SECONDARY OUTCOMES:
Diagnostic accuracy in the control set | At the end of a 2-week dermatology elective
  Mean score of the control set (number of correct answers)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Sun Yoon, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Department of Dermatology, Seoul National University Boramae Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowen JL. Educational strategies to promote clinical diagnostic reasoning. N Engl J Med. 2006 Nov 23;355(21):2217-25. doi: 10.1056/NEJMra054782. No abstract available. PMID 17124019
- [Background] Rourke L, Oberholtzer S, Chatterley T, Brassard A. Learning to detect, categorize, and identify skin lesions: a meta-analysis. JAMA Dermatol. 2015 Mar;151(3):293-301. doi: 10.1001/jamadermatol.2014.3300. PMID 25565125
- [Derived] Choi S, Oh S, Lee DH, Yoon HS. Effects of reflection and immediate feedback to improve clinical reasoning of medical students in the assessment of dermatologic conditions: a randomised controlled trial. BMC Med Educ. 2020 May 8;20(1):146. doi: 10.1186/s12909-020-02063-y. PMID 32384885